CLINICAL TRIAL: NCT02159716
Title: Phase I Study of Chimeric Antigen Receptor Modified T Cells in Patients With Mesothelin Expressing Cancers
Brief Title: CART-meso in Mesothelin Expressing Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 31213, 819826
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Pancreatic (Ductal) Adenocarcinoma; Epithelial Ovarian Cancer; Malignant Epithelial Pleural Mesothelioma
Keywords: Subjects
MeSH Terms: conditions — Adenocarcinoma; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (3):
- Metastatic Pancreatic (ductal) adenocarcinoma (PDA) (Experimental)
  Interventions: Biological: CART-meso
- Serious Epithelial Ovarian Cancer (Experimental)
  Interventions: Biological: CART-meso
- Malignant Epithelial Pleaural Mesothelioma (Experimental)
  Interventions: Biological: CART-meso

INTERVENTIONS:
Biological: CART-meso — CART-meso are autologous T cells lentivirally transduced with chimeric anti-mesothelin immunoreceptor SS1 fused to the 4-1BB and CD3ζ signaling domains.

SUMMARY:
Phase I study to establish safety and feasibility of intravenously administered lentiviral transduced CART-meso cells administered with and without cyclophosphamide in a 3+3 dose escalation design in patients with metastatic pancreatic cancer, serous epithelial ovarian cancer, or pleural mesothelioma. Dose: 1-3xE7 /mE2 (Cohort 1 and 2) and 1-3xE8 /mE2 (Cohort 3 and 4 ) CAR+ T cells by intravenous route. In the event of 2 DLTs at each dose level, we will dose deescalate by 10-fold.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cancer (one of the following):

  * Metastatic pancreatic adenocarcinoma.
  * Persistent or recurrent serous epithelial ovarian cancer or primary peritoneal carcinoma
  * Malignant pleural mesothelioma (histologically confirmed epithelial)
* Failure of at least one prior standard of care chemotherapy for advanced stage disease.
* Subjects must have measureable disease as defined by RECIST 1.1 criteria or modified RECIST criteria.
* Patients > 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy > 3 months.
* Satisfactory organ and bone marrow function as defined by the following (of note, the minimal blood counts should be in the absence of transfusion or cytokine support):

  i. Absolute neutrophil count > 1,000/μl ii. Platelets >75,000/μl iii. Hemoglobin > 9 g/dL iv. Bilirubin < 2.0x the institutional normal upper limit unless secondary to bile duct obstruction by tumor v. Creatinine < 1.5x the institutional normal upper limit vi. Albumin ≥2 vii. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 5x the institutional normal upper limit viii. Cardiac ejection fraction of >55% as measured by resting echocardiogram, with no significant pericardial effusion.
* Blood coagulation parameters: PT such that international normalized ratio (INR) is ≤ 1.5 and a PTT < 1.2 time the upper limit of normal unless the patient is therapeutically anti-coagulated for history of cancer-related thrombosis and has stable coagulation parameters.
* Ability to understand and the willingness to provide written informed consent.
* Male and Female subjects of reproductive potential agree to use approved contraceptive methods (e.g. birth control pills, barrier device, intrauterine device, abstinence) and abstain from other methods of conception during the study and for 6 months following the study cell infusion or proof of sterility.

Exclusion Criteria

* Sarcomatoid MPM histology which is known in the literature to not express mesothelin; biphasic MPM is also excluded.
* Participated in any other trial in which receipt of an investigational study drug occurred within 28 days prior to enrollment and anticipated treatment with another investigational product while on study. This refers to non-commercially approved investigational drugs different than those used in this protocol.
* Anticipated need for systemic chemotherapy within 2 weeks before apheresis and infusion of CART-meso cells.
* Active invasive cancer other than the one of the three cancers in this study. Patients with active non-invasive cancers (such as non-melanoma skin cancer, superficial cervical and bladder and prostate cancer with PSA level < 1.0) are not excluded.CART-meso in mesothelin expressing cancers
* HIV, HCV, or HBV infections
* Active autoimmune disease (including but not limited to: systemic lupus erythromatosis, Sjogren's syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, etc.) requiring immunosuppressive therapy within the past 4 weeks, with exception of thyroid replacement.
* Patients with ongoing or active infection.
* Planned concurrent treatment with systemic high dose corticosteroids. Patients may be on a stable low dose of steroids (<10mg equivalent of prednisone) for chronic respiratory conditions.
* Patients requiring supplemental oxygen therapy.
* Prior therapy with gene modified cells.
* Previous experimental therapy with SS1 moiety, murine or chimeric antibodies (human and humanized antibodies are allowed).
* History of allergy to murine proteins
* History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40)
* Any clinically significant pericardial effusion; CHF (NY Heart Association Grade II-IV) or cardiovascular condition that would preclude assessment of mesothelin induced pericarditis or that may worsen as a result of toxicities expected for this study. This determination will be made by a cardiologist.
* Any clinically significant pleural or peritoneal effusion that cannot be drained with standard approaches. An indwelling drainage device placed prior to enrollment is acceptable.
* Pregnant or breastfeeding women. Female study participants of reproductive potential must have a negative urine pregnancy test of enrollment. A serum pregnancy test will be performed within 2 weeks before infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Haas, MD, Principal Investigator — Ambramson Cancer Center of the University of Pennsylvania; Andrew Haas, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States